CLINICAL TRIAL: NCT05964816
Title: A Longitudinal Study of the Trajectory of Financial Toxicity and Its Relationship With Symptom Burden in Breast Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Yi Kuang, Principal Investigator, Fudan University
Other Study IDs: YKuang
Record Dates: First submitted 2023-07-20; First posted 2023-07-28 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Financial Toxicity
MeSH Terms: conditions — Financial Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Breast cancer has become the leading cause of global cancer incidence. With the improvement of treatment methods, some breast cancer patients have experienced different degrees of financial toxicity, which seriously affected the quality of life, treatment compliance and treatment outcomes of patients. Currently, there are some related studies on financial toxicity in breast cancer patients, but they are mainly cross-sectional studies, lacking the use of validated financial toxicity tools to measure the longitudinal change trajectory of financial toxicity. The financial toxicity of breast cancer patients may change dynamically with the treatment stage, expenditure and time, so it is necessary to conduct a rigorously designed prospective study to explore the trajectory of financial toxicity. In addition, previous studies have showed that financial toxicity may be associated with anxiety, distress, pain and overall symptom burden. However, the relevant evidence is currently limited. This study is designed as a prospective longitudinal study to explore the trajectory of financial toxicity and its influencing factors in breast cancer patients in China, and to focus on the relationship between symptom burden and financial toxicity, which will help clinicians identify potential high-risk populations, and provide a new perspective for future intervention programs.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with breast cancer and underwent surgery
* Be going to receive one or more of chemotherapy, radiotherapy, targeted therapy, endocrine therapy, and immunotherapy
* With the ability to understand and communicate in Chinese
* Provided informed consent

Exclusion Criteria:

* Illness was considered too severe for participation
* With cognitive or psychiatric disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity.
Study Population: Breast cancer patients undergoing surgery at the Fudan University Shanghai Cancer Center, the First Hospital of China Medical University, Wuhan Union Hospital and Xijing Hospital of the Fourth Military Medical University.
Sampling Method: Non-Probability Sample
Enrollment: 485 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Financial toxicity | Baseline, 3 months, 6 months, and 12 months
  Measured with the Comprehensive Scores for Financial Toxicity Based on The Patient-reported Outcome Measures (COST-PROM). The total score is 0-44, and the lower the score, the more severe financial toxicity.
Physical symptom burden | Baseline, 3 months, 6 months, and 12 months
  Measured with the Breast Cancer Prevention Trial Eight Symptom Scale (BESS), which is a 5-point severity scale. The higher the score, the more severe the physical symptom burden.
Psychological symptom burden | Baseline, 3 months, 6 months, and 12 months
  Measured with Psychologic Symptom Distress Score (PHYS) of Memorial Symptom Assessment Scale Short Form (MSAS-SF), which adopted Likert 4 scale. The higher the score, the more severe the psychological symptom burden.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Fudan University Shanghai Cancer Center, Shanghai
  - The First Hospital of China Medical University, Shenyang
  - Wuhan Union Hospital, Wuhan
  - Xijing Hospital of the Fourth Military Medical University, Xi'an

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.